CLINICAL TRIAL: NCT06705465
Title: Cross-sectorial Rehabilitation of Patients with Lung Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Camilla Balle (Other)
Responsible Party: Sponsor-Investigator, Camilla Balle, Principal investigator, phD student, Copenhagen University Hospital at Herlev
Organization: Copenhagen University Hospital at Herlev (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CBalle
Record Dates: First submitted 2024-11-22; First posted 2024-11-26 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-10

CONDITIONS: Lung Cancer Non-Small Cell Cancer (NSCLC)
Keywords: rehabilitation; cross-sectorial collaboration; video conference
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: RCT
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group: video conference (Experimental)
  Interventions: Behavioral: video conference
- No intervention (No Intervention)

INTERVENTIONS:
Behavioral: video conference — video conference
  Arms: Intervention group: video conference

SUMMARY:
Four thousand seven hundred patients are diagnosed with lung cancer in Denmark every year. Even though cigarette smoking has declined for decades a decline in lung cancer incidence is still at least a decade away. Only 16% of these patients with lung cancer started in a municipal rehabilitation program.

Aim: To investigate if the intervention "early contact conference" can facilitate acceptance of and participation in municipal rehabilitation in patients with lung cancer. Further, to investigate whether the rehabilitation improve the patients' physical ability and quality of life.

Thirteen municipalities from Region Hovedstaden have agreed to participate in this cluster randomized controlled trial. The intervention will focus on creating early contact between the Department of Oncology and the municipalities. The conference call will be planned when the patient is at the hospital for the second systemic treatment and a written status will be sent to the GP after the conference video call so that hospital, municipality, and GP will all have the newest knowledge about the patient's general condition

The intervention will be easy to implement in clinical practice afterwards if it is a success and the cost of the intervention is low.

DETAILED DESCRIPTION:
Cross-sectorial rehabilitation of patients with lung cancer - A cluster randomized controlled trial

Background Currently, approximately 4,700 patients are diagnosed with lung cancer annually in Denmark, with equal distribution between men and women. The average age at the time of diagnosis is 69 years, and the majority of patients are smokers or former smokers, with a high incidence of age- and smoking-related comorbidities. Lung cancer is divided into small cell lung cancer (SCLC) and non-small cell lung cancer (NSCLC). Patients with very small tumors are offered surgery. Otherwise, treatment of localized disease consists of systemic treatment in combination with radiotherapy. Patients with disseminated disease are primarily treated with palliative chemotherapy, targeted treatment or immunotherapy.

The standard program in 2024 for rehabilitation and palliation of patients with cancer in Denmark is a nationwide, multidisciplinary approach defining the roles and the responsibilities of the hospital, municipality and general practice. At the hospital the patients are informed about possible rehabilitation and referred to the municipalities. This is done through a "needs assessment". A needs assessment must be offered at the beginning of treatment, at the end, and during follow-up care, as well as when there are changes in treatment or disease status. This, to ensure that all patients are offered an evaluation of current challenges and needs for support to maintain or restore daily life.

Continuity of care across sectors is a major challenge for healthcare systems. This affects patients with chronic disorders, such as cancer. It is difficult to motivate patients with lung cancer for rehabilitation and exercise, although, they often have many physical challenges, multiple comorbidities and concurrent symptoms. Both patients with lung cancer treated with a curative intent and those with advanced disease can experience fatigue, shortness of breath, pain, cough, depression, weight loss, and decreased muscle strength. Patients often avoid behaviors that produce symptoms and maintain an inactive pattern that exacerbates these symptoms.

A Danish survey, encompassing over 3,000 patients with cancer, reveals that 58% of the patients required support from the municipality. Additionally, 74% of the patients report discomfort that significantly impacts their daily lives due to the cancer and/or treatment. The survey also indicates that many cancer patients are not informed about rehabilitation. Specifically, 52% of patients report that a health professional has not discussed how their general practitioner can assist them with their cancer-related needs, and 40% report that they have not been informed about the support available from the municipality. Thus, data from Department of Oncology, Herlev and Gentofte Hospital's record system shows that only 16% of patients with lung cancer started rehabilitation in 2022. So there seems to be a major communication gap between the sectors in the Danish health care system.

Various shared care models have been developed in the field of cancer, primarily involving the general practitioner (GP) and the oncologist. Multidisciplinary video consultations are one method to improve coherence and coordination of care for patients with cancer. Seeing each other is essential for building and establishing professional relationships and can be accomplished through video. In a Danish study including patients in a shared video consultation with the GP and the oncologist;, 90% of the included patients, expressed that it was beneficial to have both doctors present. Furthermore, studies have highlighted how video consultations can contribute to effective and inclusive communication, and facilitate a feeling of security, trust and relationship building although sitting apart.

Hypothesis and aims We hypothesize that many patients with lung cancer have unmet rehabilitation needs and that an early video conference with the patient, specialist nurse and the coordinator from the municipality - the early contact conference - will increase the percentage of patients accepting rehabilitation.

The aim is to investigate if the intervention "early contact conference" facilitates acceptance and start of participation in municipal rehabilitation in patients with NSCLC undergoing systemic cancer treatment.

Research question

Primary outcome:

• Will an "early contact conference" with the primary sector increase the number of patients with NSCLC starting rehabilitation in the municipality?

Secondary outcomes:

* Will an "early contact conference" contribute to more patients maintaining municipal rehabilitation?
* Will Quality of life (Qol) and physical functions increase in patients receiving rehabilitation compared to patients who do not attend rehabilitation?
* Will an "early contact conference" decrease the numbers and duration of hospitalizations? Our definition of maintaining rehabilitation: the patient attends three or more appointments or ≥ 50% of planned intervention.

Design A cluster randomized controlled trial (RCT). Thirteen municipalities from Region Hovedstaden have agreed to participate in the RCT. Three municipalities have declined. The thirteen municipalities will be randomized to be either intervention or control municipalities. The randomization of the municipalities will be stratified according to the socioeconomic status of the municipality and to the number of patients the clinic receives from the individual municipality.

Methods Population Participants in this project are men and women ≥ 18 years of age who are receiving first line systemic treatment for NSCLC at the Department of Oncology, Herlev and Gentofte Hospital. Only patients who cannot speak, understand, and/or read Danish or who are judged to be cognitively/psychologically unfit to give consent to participate in the project will be excluded. Patients who are resident in a non-participating municipality will also be excluded. The reason for excluding patients will be registered.

Recruitment of participants The treatment course for patients with lung cancer starts with the patient attending a medical consultation in the clinic, where the treatment plan is reviewed. On the 2nd day, the patient comes in for the first consultation with the nurse, where the oncologist's consultation is followed up. On the 3rd day, the patient starts treatment (chemotherapy and/or immunotherapy).

Eligible participants for the project are identified by nurses in the lung cancer team at the Department of Oncology, Herlev and Gentofte hospital and are informed about the project at the first nurse interview on the 2nd day. If the patient accepts to participate in the project, the patient will sign a consent form. If the patient wants to have a longer period of reflection regarding participation, the patient will be asked again at the next visit to the clinic (i.e. the 3rd day before the patient starts the first systemic treatment).

Intervention The participating municipalities are randomized in advance. Thus, the nurse knows beforehand which group the patient belongs to.

Intervention group Investigating the feasibility of rehabilitation initiation by a video conference with the patient and the relevant healthcare persons from the hospital and the municipality. The intervention will focus on creating early contact with the primary sector. The conference call will be planned when the patient is at the hospital for the second systemic treatment, or as close to this treatment as possible (2-6 weeks from first systemic treatment). A written status will be sent to the GP after the conference video call so that hospital, municipality, and GP will all have the newest knowledge about the patient's general condition. If the patient does not have any rehabilitation needs at the time of the conference call, the coordinator from the municipality will call the patient 4-5 weeks later to follow up and check if the patients need for rehabilitation have changed.

Control group The patients will have a needs assessment with the nurse from the clinic at their second day in the clinic, i.e., the day before their first systemic treatment.

Data collection

The following data will be collected from both groups:

Physical function and QoL will be measured at baseline, 1 month, 3 months and 6 months after initiation of systemic treatment. The physical tests will be performed by the nurses in the clinic. Physical function will be measured with the 30-second chair stand test (30s-CST) and hand grip strength test. The hand grip strength test will only be performed at baseline. The European Organisation for Research and Treatment of Cancer (EORTC) QLQ-C30 will be used for measuring QoL. Data on the participants' cancer-specific and general health status (age, sex, comorbidity, cancer stage, treatment purpose, type of systemic treatment, Eastern Cooperative Oncology Group Performance Status (ECOG PS)) will be obtained from the electronic medical record. The patient must fill out a short questionnaire about living status and level of education at the baseline test. The patient's weight will be recorded at each of the four test sessions. Hospitalizations under the treatment will also be recorded.

Primary endpoint:

The primary endpoint is the number of patients who attend rehabilitation once or more.

Secondary endpoints:

* The number of referrals to municipal rehabilitation. The proportion of patients receiving a referral will be compared between the municipalities in the intervention group and the control group
* The attendance and compliance of rehabilitation will be obtained from the municipal records
* Changes in QoL and 30s-CST within groups and between groups
* Numbers and duration of hospitalizations within groups and between groups
* Changes in weight within groups and between groups

The EORTC QLQ-C30 Assess quality of life (QoL). The EORTC QLQ-C30 contains 30 questions and is designed specifically to assess the QoL of patients with cancer. It has been translated and validated into over 100 languages, including Danish, - and is widely used.

The 30-second chair stand test The 30-second chair stand test (30s-CTS) measures how many times a person can get up from a chair in 30 seconds. The changes in 30s-CST will be compared between the intervention and control groups. The purpose of the test is to examine the strength and function of the lower extremity. This test is valid and reliable for assessing lower extremity strength and function in healthy older adults. The test result is considered to give an expression of functional independence. Decreased strength is a predictor of falls.

The hand grip strength test The handgrip strength test (HST) measures physical function of the upper body and will be measured using a hand-held dynamometer. The best of three attempts performed with the dominant hand will be used as test score. The handgrip strength is independently associated with functional capacity, QoL and survival in patients with advanced cancer.

Sample size and power calculation The sample size calculation is based on that 16% of the lung cancer patients are participating in a rehabilitation intervention after discharge from the hospital. In this cluster randomized trial, we expect an increase to 32% in the intervention group, and assuming a mean of 10 participants in each cluster (municipality), accepting a variation on cluster size of 0.5. A correlation of 0.1 (rho) within clusters is expected and with a power of 80% (beta) and level of significance on 0.05 (alpha) five clusters is needed in each group with 50 participants. Including 65 participants in each group will allow a dropout rate of 20%.

Statistical analyses Proportion of referrals and proportion of patients attending and completing rehabilitation in the two groups will be compared using the χ2-test. Baseline characteristics will be presented as medians and interquartile ranges (IQRs) for quantitative variables and as numbers and percentages for categorical variables. Data on physical tests will be presented as means and standard deviation (SD) or medians and IQRs, as appropriate. All tests will be two-sided and performed on a significance level of 0.05.

Feasibility From the electronical medical record, we know how many new patients with NSCLC that starts systemic treatment at the Department of Oncology, Herlev and Gentofte Hospital each year. We know how many patients we can except to receive from each participating municipality. Based on these numbers, we except to include the desired number of 130 participants (65 in each group) in approximately 1½-2 years.

Cross-sectorial cooperation In this cluster RCT the cross-sectorial cooperation is the key to making the intervention a success. If the intervention does not make sense for both sectors, then it will not make a difference for the patients. Therefore, the planning of the intervention is done in close cooperation between the sectors. By having two representatives from the municipalities in the project group, we hope to be able to consider everyone's needs and schedules.

Ethical considerations The project description has been submitted to the Scientific Ethics Committee and is assessed as not subject to notification (re. F-24037191). All personal data will be kept strictly confidential in a REDCap database affiliated to the research project and in accordance with the rules of the General Data Protection Regulation (GDPR) (EU) 2016/679 and Danish Law on Data Protection (Databeskyttelsesloven). The trial is registered at "Region Hovedstadens Videnscenter for Dataanmeldelser". All potential participants will be provided with full and adequate verbal and written information about the project and will have the right to ask questions about the study. Each patient will be informed about their personal rights when entering the study. It is emphasized that participation in the study is voluntary, and that any included patients at any given time can cancel participation in the study.

Relevance and perspective The intervention is implementable in the clinic and can be used for patients with other cancer diagnosis. It can also be a relevant tool in other course programs for chronic illness (e.g. diabetes, cardiovascular diseases) because the referral to the municipality is similar.

Dissemination The study results will be presented in a peer reviewed journal and at local, national, and international conferences. The results will also be shared with health professionals from both sectors in Region Hovedstaden through dialogue meetings. A meeting form that is already establish between the Department of Oncology, Herlev and Gentofte Hospital and the municipalities. The general practitioners will also be invited.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with NSCLC
* 1. line systemic treatment

Exclusion Criteria:

* cannot speak, understand, and/or read Danish
* cognitive/psychologically unfit to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2024-10-07 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Early contact conference | 6 months after treatment start
  • Will an "early contact conference" with the primary sector increase the number of patients with NSCLC starting rehabilitation in the municipality?

SECONDARY OUTCOMES:
Quality of life | EORTC-C30 baseline, 3 weeks, 9 weeks, 6 months
  • Will Quality of life (Qol) and physical functions increase in patients receiving rehabilitation compared to patients who do not attend rehabilitation? The EORTC QLQ-C30 Measurement of QoL: The EORTC QLQ-C30 30 questions and is designed specifically to assess the QoL of patients with cancer.
  Measurement of physical function: The 30-second chair stand test (30s-CTS) measures how many times a person can get up from a chair in 30 seconds.

CONTACTS AND LOCATIONS:
Locations (1):
- Herlev and Gentofte Hospital, Herlev, Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No